CLINICAL TRIAL: NCT07297251
Title: Assessment of Temporomandibular Joint Mobility With Different Head Postures. Analysis of the Influence of Selected Manual Therapy Techniques on Temporomandibular Joint Mobility and Head Posture.
Brief Title: Temporomandibular Joints Mobility and Head Posture: Influence of Manual Therapy and Exercises in Dental Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Resolution No. 5-II/2024
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular joint; range of motion; cervical spine; kinematic; manual therapy; exercices
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual therapy (Other): Manual therapy, exercises
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — 1. Performance of 2 manual therapy techniques immediately following the participant's initial examination. The participant remains secured in the device. The examiner performs manual therapy on each temporomandibular joint (TMJ) sequentially. The following procedures are performed consecutively: 6 sec. of Grade II distraction (traction) according to F. Kaltenborn on the TMJ, repeated 6 times; 6 seconds of Grade II lateral glide on the TMJ, repeated 6 times. Following the completed physiotherapy intervention, the digital axiograph examination is performed again. A comparative analysis of the performed examinations will be conducted
  2. Instruction on homework exercises performed by the patient. The exercises are performed 6 times per day, each in a series of 6 repetitions, for a period of 4 to 6 weeks. They include: a) Head flexion in the cranio-cervical joint - Standing position near a door frame; the patient performs maximum head flexion while simultaneously resting the occiput against

SUMMARY:
Goal: This clinical study aims to investigate how the range of motion of the temporomandibular joints (TMJ) changes in relation to the patient's head posture. Furthermore, we will assess the efficacy of a specific physiotherapy program in improving TMJ mobility and influencing head alignment in patients undergoing orthodontic treatment or prosthetic reconstruction.

Scope: The project will evaluate TMJ function and head alignment in orthodontic or prosthetic patients aged 11-65. The core focus is to analyze the correlation between head posture and TMJ mobility and to measure changes in these parameters before and after the manual physiotherapy intervention.

DETAILED DESCRIPTION:
This study is designed to address the complex and often debated biomechanical relationship between craniocervical posture (head-to-neck alignment) and the function of the temporomandibular joint (TMJ). Clinical evidence suggests a strong link between forward head posture and temporomandibular disorders (TMDs). However, objective quantification of TMJ mobility changes induced purely by varying head position remains insufficiently documented. This trial seeks to establish a clear, quantifiable relationship and evaluate a targeted manual therapy intervention designed to optimize both head posture and TMJ function.

Objectives and Specific Aims

The overarching goal is to determine the dependence of temporomandibular joint mobility on the patient's head posture relative to the body, and to assess the impact of a defined physiotherapy program on these parameters.

Specific Aims include:

Functional Assessment: To perform a baseline functional evaluation of the TMJ in patients (aged 11 to 65) who are undergoing orthodontic treatment or require prosthetic reconstruction.

Postural Measurement: To objectively assess the resting position of the head relative to the cervical spine in the context of the current dental state (orthodontic appliance use or pre-prosthetic condition).

Correlational Analysis: To establish and quantify the relationship between measured TMJ mobility (e.g., maximum mouth opening, lateral excursion) and various head postures (e.g., neutral, forward, retracted).

Intervention Efficacy: To conduct a detailed pre- and post-intervention functional evaluation of the TMJ and head posture following the completion of a defined physiotherapy program for all eligible participants.

Change Quantification: To determine the magnitude and direction of changes in both TMJ mobility and head alignment resulting from the implemented physiotherapy protocol.

Study Design and Methodology

This will be a multi-center, prospective, interventional study with a pre- and post-intervention assessment design. Participants will be recruited from dental and physiotherapy clinics.

Participants: The study population will include patients aged 11 to 65 years who are either undergoing active orthodontic treatment or are scheduled for complex prosthetic reconstruction.

Intervention: The intervention group will receive a standardized program of manual physiotherapy and exercises. The program will be delivered over a fixed duration (e.g., 6 weeks, 12 sessions).

Outcome Measurement: All measurements will be performed at baseline (Pre-Intervention) and upon completion of the physiotherapy program (Post-Intervention).

TMJ Mobility: Measured objectively using a Jaw Motion Analyzer Axiograph

Maximum unassisted and assisted mouth opening (MIO/MMO), left and right lateral excursions, protrusion/retrusion.

Head Posture: Measured objectively using established clinical photography methods and.CROM device

Duration and Follow-up

The total duration of the study is anticipated to be 3 years for recruitment and data collection. Each participant's active involvement will span [e.g., 8 weeks], encompassing baseline assessment, the physiotherapy period, and the final assessment. No long-term follow-up beyond the final assessment is currently planned.

Data Analysis

Statistical analysis will employ methods appropriate for repeated measures. Primary analysis will focus on calculating Pearson's correlation coefficients to assess the relationship between initial head posture and TMJ mobility. Secondary analysis will utilize paired t-tests (or non-parametric equivalents) to determine the statistical significance of changes in TMJ mobility and head posture between the pre- and post-intervention phases. (Include specific statistical software, e.g., SPSS or R, if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 11 to 13 years with a confirmed occlusion class (Class I, II, or III) with parental/legal guardian consent.
* Patients aged 13 to 17 years with personal assent and parental/legal guardian consent.
* Adult patients (up to 65 years of age) who have provided informed consent.

Exclusion Criteria:

* Inability to perform required study tests or procedures.
* Positive safety tests indicating contraindications to manual intervention.
* History of surgeries or trauma to the maxillofacial region.
* Genetic defects or neurological disorders.
* Current orthodontic treatment with fixed appliances.
* Current splint therapy.
* Pregnancy.
* Lack of consent from a parent or legal guardian (for minors).
* Lack of cooperation from the participant (especially children).

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
CROM device | Baseline and after 1 and 2 months
  Cervical spine movements
JMA (Jaw Motion Analyzer) Axiograph | Baseline and after 1 and 2 months
  TMJ movements

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaczmarek B, Kaczmarek L, Mysliwiec A, Lipowicz A, Dowgierd K. Kinematic Relationship Between Temporomandibular and Cervical Spine Joints. J Oral Rehabil. 2025 Sep;52(9):1496-1504. doi: 10.1111/joor.14015. Epub 2025 May 9. PMID 40346746